CLINICAL TRIAL: NCT06696911
Title: Combined Effects of Motor Imagery and Core Stability Exercises on Trunk Control, Balance and Quality of Sleep in Stroke Patients
Brief Title: Combined Effects of Motor Imagery and Core Stability Exercises in Stroke Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0239
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Stroke; Core Stability Exercises; Motor Imagery; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stability Exercises and Motor Imagery (Experimental): Core stability exercises are voluntary movements designed to maintain the balance, functional mobility, gait, fear of falling, and anticipatory postural adjustment among stroke survivors. Motor perception or motor imagery (MI) is a mental task that involves visualizing a physical movement without actually doing the action
  Interventions: Procedure: Core stability Exercises; Procedure: Motor Imagery
- Core Stability Exercises (Active Comparator): Core stability exercises are voluntary movements designed to maintain the balance, functional mobility, gait, fear of falling, and anticipatory postural adjustment among stroke survivors.
  Interventions: Procedure: Motor Imagery

INTERVENTIONS:
Procedure: Core stability Exercises — The exercises have been divided into three difficulty categories based on the level of difficulty.
  Level I: When the patients were unable to sit independently, level I core stability therapy was administered. First-level exercises were done in a supine position on a plinth. The workout program mostly included side bridging movements, leg crosses, one-leg curl-ups, and straight and diagonal reaching activities. Patients can move to level once they can sit on a plinth edge unsupported for one minute while flexing their knees and hips to 90 degrees.
  Level II: Exercises included straight-arm curl-ups, diagonal-arm curl-ups, and arm curl-ups with the arms crossed. The patient will go to stage three once they can sit on an unstable surface for thirty seconds.
  Level III: Using a physio ball, the exercises were done while seated. The exercises performed with the ball consisted push-ups, bird dog, side Bridge, abdominal curl-ups, and bridge movements
  Arms: Core Stability Exercises and Motor Imagery
Procedure: Motor Imagery — The motor imagery program will be performed in three steps. STEP 1 Subjects will be instructed to watch the video provided and recorded by investigator. Two types of videos will be available to watch. One recording normal movements and the other film will contain recording the patient movements. Patient will be asked to watch the video and analyze the differences.
  STEP 2 In next step participants will be asked to close the eyes to focus and then to imagine how they are doing task they had previously observed 10 times.
  STEP 3 Participants will be than instructed to carry out the task in verbal commands given whenever necessary. During the recall process components of movement deviating from normal will be emphasized. The difficulty level of activities and the analysis of movement components will be increased gradually according to the patient's capacity.

SUMMARY:
This research explores the combined effects of motor imagery and core stability exercises on trunk control, balance, and sleep quality in stroke recovery, addressing Pakistan's unique healthcare challenges. By enhancing neuroplasticity, core strength, and physical function, these interventions aim to improve mobility, independence, and overall quality of life for stroke survivors, while addressing common sleep disturbances.

DETAILED DESCRIPTION:
Stroke patients can benefit from motor imagery and mirror therapy, which are easy to perform anytime and anywhere at their convenience. Integrating motor imagery training with task-specific training leads to greater improvements in sit-to-stand performance compared to task-specific training alone. Core exercises, whether performed alone or combined with other therapies, have been shown to influence trunk performance in stroke patients compared to traditional training. Patients who have had strokes can benefit from rehabilitation training that focuses on strengthening their core muscles. This is likely because it thickens the transverse abdominis muscle. Post-stroke patients were able to regain their motor function and sense of independence with the use of motor imagery as an additional resource. It has been shown to be an effective therapeutic strategy for this particular patient population. More than with routine physiotherapy, core stability exercises on both stable and unstable support surfaces improve ambulatory stroke patients' trunk control, core muscular strength, standing weight-bearing symmetry, and balance confidence. Combined action observation and motor imagery therapy may be helpful for neurorehabilitation in chronic stroke survivors when physical practice is not appropriate. Compared to standard physical treatment alone, core stability exercise and conventional physical therapy has demonstrated better outcomes in trunk control and balance.

The combination of motor imagery and core stability exercises remains underexplored in stroke rehabilitation, leaving a significant knowledge gap about their synergistic potential. Investigating their combined effects could offer innovative strategies to improve trunk control, balance, and sleep quality, paving the way for more comprehensive and effective post-stroke treatment programs.

ELIGIBILITY:
Inclusion Criteria: Adults aged 40-65 years.

* Diagnosed with stroke (ischemic or hemorrhagic) within the last 6 months to 2 years.
* Hemiplegic Patient
* Having MMSE score ≥ 24
* Experiencing balance impairments on BBS 21-40
* Having sleep disturbances on PSQI 15-21.
* Willing to provide informed consent.

Exclusion Criteria: Severe cognitive impairments (e.g., severe dementia).

* Other neurological or musculoskeletal conditions affecting balance.
* Severe cardiovascular or respiratory conditions contraindicating exercise.
* Participation in another clinical trial within the past 3 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
• Berg Balance Scale ( BBS) | 12th week
  The Berg Balance Scale evaluates changes in static balance over time .Each item is a 5-point ordinal scale ranging from 0 to 4, with 0 indicating lowest level of function and 4 indicating highest level of function. It has 14 items and the maximum score is 56, higher the score, the better the balance function, while the lower the score, the worse the balance function.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd, Principal Investigator — Riphah International University
Locations (1):
- Well Versed Physio Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kashif M, Ahmad A, Bandpei MAM, Gilani SA, Hanif A, Iram H. Combined effects of virtual reality techniques and motor imagery on balance, motor function and activities of daily living in patients with Parkinson's disease: a randomized controlled trial. BMC Geriatr. 2022 Apr 30;22(1):381. doi: 10.1186/s12877-022-03035-1. PMID 35488213
- [Background] Niu S, Liu X, Wu Q, Ma J, Wu S, Zeng L, Shi Y. Sleep Quality and Cognitive Function after Stroke: The Mediating Roles of Depression and Anxiety Symptoms. Int J Environ Res Public Health. 2023 Jan 29;20(3):2410. doi: 10.3390/ijerph20032410. PMID 36767777
- [Background] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Background] Miyata K, Tamura S, Kobayashi S, Takeda R, Iwamoto H. Berg Balance Scale is a Valid Measure for Plan Interventions and for Assessing Changes in Postural Balance in Patients with Stroke. J Rehabil Med. 2022 Dec 9;54:jrm00359. doi: 10.2340/jrm.v54.4443. PMID 36484715
- [Background] Park M, Seok H, Kim SH, Noh K, Lee SY. Comparison Between Neuromuscular Electrical Stimulation to Abdominal and Back Muscles on Postural Balance in Post-stroke Hemiplegic Patients. Ann Rehabil Med. 2018 Oct;42(5):652-659. doi: 10.5535/arm.2018.42.5.652. Epub 2018 Oct 31. PMID 30404414
- [Background] Liu W, Cheng X, Rao J, Yu J, Lin Z, Wang Y, Wang L, Li D, Liu L, Gao R. Motor imagery therapy improved upper limb motor function in stroke patients with hemiplegia by increasing functional connectivity of sensorimotor and cognitive networks. Front Hum Neurosci. 2024 Feb 19;18:1295859. doi: 10.3389/fnhum.2024.1295859. eCollection 2024. PMID 38439937
- [Background] Binks JA, Emerson JR, Scott MW, Wilson C, van Schaik P, Eaves DL. Enhancing upper-limb neurorehabilitation in chronic stroke survivors using combined action observation and motor imagery therapy. Front Neurol. 2023 Mar 2;14:1097422. doi: 10.3389/fneur.2023.1097422. eCollection 2023. PMID 36937513
- [Background] Karthikbabu S, Ganesan S, Ellajosyula R, Solomon JM, Kedambadi RC, Mahabala C. Core Stability Exercises Yield Multiple Benefits for Patients With Chronic Stroke: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Apr 1;101(4):314-323. doi: 10.1097/PHM.0000000000001794. PMID 34001840
- [Background] Chen X, Gan Z, Tian W, Lv Y. Effects of rehabilitation training of core muscle stability on stroke patients with hemiplegia. Pak J Med Sci. 2020 Mar-Apr;36(3):461-466. doi: 10.12669/pjms.36.3.1466. PMID 32292453
- [Background] Cabrera-Martos I, Ortiz-Rubio A, Torres-Sanchez I, Lopez-Lopez L, Jarrar M, Valenza MC. The Effectiveness of Core Exercising for Postural Control in Patients with Stroke: A Systematic Review and Meta-Analysis. PM R. 2020 Nov;12(11):1157-1168. doi: 10.1002/pmrj.12330. Epub 2020 Feb 17. PMID 31950672
- [Background] Lee SA, Cha HG. The effect of motor imagery and mirror therapy on upper extremity function according to the level of cognition in stroke patients. Int J Rehabil Res. 2019 Dec;42(4):330-336. doi: 10.1097/MRR.0000000000000366. PMID 31425348
- [Background] Ma ZZ, Wu JJ, Hua XY, Zheng MX, Xing XX, Ma J, Li SS, Shan CL, Xu JG. Brain Function and Upper Limb Deficit in Stroke With Motor Execution and Imagery: A Cross-Sectional Functional Magnetic Resonance Imaging Study. Front Neurosci. 2022 May 19;16:806406. doi: 10.3389/fnins.2022.806406. eCollection 2022. PMID 35663563
- [Background] Jeffers MS, Pittman AC, Kendzerska T, Corbett D, Hayward KS, Chen Y. Self-reported sleep disturbances among people who have had a stroke: a cross-sectional analysis. CMAJ. 2023 Mar 14;195(10):E354-E362. doi: 10.1503/cmaj.221063. PMID 36918185
- [Background] Iddagoda MT, Inderjeeth CA, Chan K, Raymond WD. Post-stroke sleep disturbances and rehabilitation outcomes: a prospective cohort study. Intern Med J. 2020 Feb;50(2):208-213. doi: 10.1111/imj.14372. PMID 31111660
- [Background] Zhang Y, Wang C, Yang J, Qiao L, Xu Y, Yu L, Wang J, Ni W, Wang Y, Yao Y, Yong Z, Ding S. Comparing the Effects of Short-Term Liuzijue Exercise and Core Stability Training on Balance Function in Patients Recovering From Stroke: A Pilot Randomized Controlled Trial. Front Neurol. 2022 Feb 10;13:748754. doi: 10.3389/fneur.2022.748754. eCollection 2022. PMID 35242094
- [Background] Khallaf ME. Effect of Task-Specific Training on Trunk Control and Balance in Patients with Subacute Stroke. Neurol Res Int. 2020 Nov 17;2020:5090193. doi: 10.1155/2020/5090193. eCollection 2020. PMID 33294224
- [Background] Cabanas-Valdes R, Bagur-Calafat C, Girabent-Farres M, Caballero-Gomez FM, Hernandez-Valino M, Urrutia Cuchi G. The effect of additional core stability exercises on improving dynamic sitting balance and trunk control for subacute stroke patients: a randomized controlled trial. Clin Rehabil. 2016 Oct;30(10):1024-1033. doi: 10.1177/0269215515609414. Epub 2015 Oct 8. PMID 26451007
- [Background] Sonmez I, Karasel S. Poor Sleep Quality I Related to Impaired Functional Status Following Stroke. J Stroke Cerebrovasc Dis. 2019 Nov;28(11):104349. doi: 10.1016/j.jstrokecerebrovasdis.2019.104349. Epub 2019 Sep 3. PMID 31492629
- [Background] Monteiro KB, Cardoso MDS, Cabral VRDC, Santos AOBD, Silva PSD, Castro JBP, Vale RGS. Effects of Motor Imagery as a Complementary Resource on the Rehabilitation of Stroke Patients: A Meta-Analysis of Randomized Trials. J Stroke Cerebrovasc Dis. 2021 Aug;30(8):105876. doi: 10.1016/j.jstrokecerebrovasdis.2021.105876. Epub 2021 May 25. PMID 34049014
- [Background] Khazaei S, Ayubi E, Khazaei M, Khazaei M, Afrookhteh G. Sleep Quality and Related Determinants among Stroke Patients: A Cross-Sectional Study. Iran J Psychiatry. 2022 Jan;17(1):84-90. doi: 10.18502/ijps.v17i1.8052. PMID 35480131
- [Background] Xiao M, Huang G, Feng L, Luan X, Wang Q, Ren W, Chen S, He J. Impact of sleep quality on post-stroke anxiety in stroke patients. Brain Behav. 2020 Dec;10(12):e01716. doi: 10.1002/brb3.1716. Epub 2020 Nov 3. PMID 33140545